CLINICAL TRIAL: NCT01378234
Title: The Impact of a Social Work Driven Transitional Care Model on Health Outcomes for At-Risk Older Adults
Brief Title: Enhanced Discharge Planning Program -- Prospective
Acronym: EDPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Robyn Golden, Associate Vice President, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 08121903-IRB02
Record Dates: First submitted 2011-06-17; First posted 2011-06-22 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Patient Admission; Patient Discharge
MeSH Terms: interventions — 2-ethylidene-1,5-dimethyl-3,3-diphenylpyrrolidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EDPP Intervention (Experimental): Receive EDPP transitional care intervention from social worker upon hospital discharge
  Interventions: Behavioral: Enhanced Discharge Planning Program transitional care
- Usual Care (No Intervention): Receive usual care upon hospital discharge

INTERVENTIONS:
Behavioral: Enhanced Discharge Planning Program transitional care — Enhanced Discharge Planning Program (EDPP) provides telephonic short-term post-discharge social work services that assess and intervene from a biopsychosocial perspective for at-risk older adults returning home after an inpatient hospitalization. EDPP follows a four-step process to with three guiding tasks to reach the goal of preventing avoidable adverse events post-discharge:
  1. Ensure patients understand the discharge plan of care and receive recommended services while screening for unidentified medical or social needs
  2. Connect patients to outpatient health services (ex: home health, in-home services, dialysis, radiology, laboratory services, specialty care) with particular emphasis on the first physician follow-up appointment
  3. Supporting caregivers to reduce stress and burden
  Other Names: EDPP
  Arms: EDPP Intervention

SUMMARY:
The Enhanced Discharge Planning Program (EDPP) is an intervention designed to help older adults safely transition to the community after discharge. This is achieved through telephonic care coordination facilitated by social workers. EDPP social workers ensure full implementation of the discharge plan, assist with coordinating community resources and follow-up appointments, and intervene around other issues that may arise as a result of a complex transition.

The EDPP intervention is currently being offered to some older adult patients discharged from Rush University Medical Center. Case managers refer older adult patients on selected units who they believe may be at risk for adverse events post-discharge. While this service is being provided to patients, it has not yet been formally evaluated. This randomized controlled trial will provide data necessary for a more rigorous evaluation of the efficacy of this intervention.

DETAILED DESCRIPTION:
The Enhanced Discharge Planning Program (EDPP) is an intervention designed to help older adults safely transition to the community after discharge. This is achieved through telephonic care coordination facilitated by social workers. EDPP social workers ensure full implementation of the discharge plan, assist with coordinating community resources and follow-up appointments, and intervene around other issues that may arise as a result of a complex transition.

The EDPP intervention is currently being offered to some older adult patients discharged from Rush University Medical Center. Case managers refer older adult patients on selected units who they believe may be at risk for adverse events post-discharge. While this service is being provided to patients, it has not yet been formally evaluated. This randomized controlled trial will provide data necessary for a more rigorous evaluation of the efficacy of this intervention.

Research Process

1. Rush University Medical Center inpatients receive the Enhanced Discharge Planning Program information sheet in the Rush patient education packet.

   All Rush inpatients will receive an informational sheet about the EDPP study, with an exception of pediatric and labor/delivery inpatients. The sheet will be included in the patient education packets distributed by Rush. This will make patients aware of the EDPP program before they leave the hospital and prepare them for a call once they return home.
2. Eligible patients are referred to the Enhanced Discharge Planning Program at their point of discharge via an electronic referral report through Epic.

   EDPP receives an electronic referral report of all patients meeting the specified referral criteria. Referral is dependent on discharge data recorded by Rush nurses and case managers in the Epic electronic medical record and generated at the point of discharge. The electronic system ensures a streamlined, standardized referral process by creating an automatic referral based upon documentation completed as part of nurse's and case manager's typical workflow. An anticipated 720 patients will be electronically referred during the duration of the study.
3. The Enhanced Discharge Planning Program project coordinator receives the daily referral report and inputs patients into the block randomization scheme.

   The project coordinator will input referrals into the existing block randomization scheme after receiving the electronic report at the beginning of the day. Referrals will be copied into the scheme in the same order as reported - sorted by episode number - to reduce bias. Patients assigned to the intervention group will be forwarded to the EDPP social workers. The usual care group will be managed by the project coordinator and student interns under her direct supervision.
4. The Enhanced Discharge Planning Program social worker contacts the intervention group to provide clinical care and obtain consent.

ELIGIBILITY:
Inclusion Criteria:

* Must meet all the following criteria:
* Aged 65+
* English speaking
* Returning home after discharge
* 7+ medication prescribed
* Must also meet one additional criterion:
* Lives alone
* Without a source of emotional support
* Without a support system for care in place
* Discharged with a service referral
* High risk for falls
* Inpatient hospitalization within 12 months
* Identified in depth psychosocial need
* High risk medication prescribed

Exclusion Criteria:

* Primary diagnosis of transplant
* Non-English speaking
* Discharged to a facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 740 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Readmissions | 30 days
  Readmission to hospital within 30 days after index discharge date
Readmissions | 60 days
  Readmission to hospital within 60 days of index discharge date
Readmissions | 90 days
  Readmission to hospital within 90 days of index discharge date
Readmissions | 180 days
  Readmission to hospital within 180 days of index discharge date

SECONDARY OUTCOMES:
Stress | 30 days
  Patient and caregiver stress, self-reported
Physician follow-up | 30 days
  Appointment made, kept with doctor
Mortality | 30 days
  patient's Mortality will be monitored and documented.
Patient needs | 30 days
  Audit of problems detected post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Golden, LCSW, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States